CLINICAL TRIAL: NCT00716807
Title: Modeling Kappa Opioid Analgesic Mechanisms in Chronic Orofacial Pain Disorders
Brief Title: Efficacy of Nalbuphine and Naloxone Administered as Nose Sprays in the Treatment of Orofacial Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit a sufficient number of subjects.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NIH/NIDCR R01 DE018526-1; 1R01DE018526-01 (NIH)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2013-10

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Burning Mouth Syndrome
Keywords: BMS; TMD
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Burning Mouth Syndrome | interventions — Nalbuphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TMD 1 (Experimental)
  Interventions: Drug: nalbuphine plus naloxone
- TMD 2 (Placebo Comparator)
  Interventions: Drug: nalbuphine plus placebo
- BMS 1 (Experimental)
  Interventions: Drug: nalbuphine plus naloxone
- BMS 2 (Placebo Comparator)
  Interventions: Drug: nalbuphine plus placebo

INTERVENTIONS:
Drug: nalbuphine plus naloxone — Patient group: temporomandibular disorders. Nalbuphine 5 mg administered by nasal spray (one time only). Naloxone 0.4 mg administered by nasal spray (one time only).
  Arms: TMD 1
Drug: nalbuphine plus placebo — Patient group: temporomandibular disorders. Nalbuphine 5 mg administered by nasal spray (one time only). Placebo (naloxone vehicle) administered by nasal spray (one time only).
  Arms: TMD 2
Drug: nalbuphine plus naloxone — Patient group: burning mouth syndrome. Nalbuphine 5 mg administered by nasal spray (one time only). Naloxone 0.4 mg administered by nasal spray (one time only).
  Arms: BMS 1
Drug: nalbuphine plus placebo — Patient group: Burning mouth syndrome. Nalbuphine 5 mg administered by nasal spray (one time only). Placebo (naloxone vehicle) administered by nasal spray (one time only).
  Arms: BMS 2

SUMMARY:
Patients with chronic masticatory muscle pain (i.e., pain greater than three months) or patients with burning mouth syndrome participate in this study. The aim of the study is to compare the pain killing effectiveness of nalbuphine, a narcotic pain killer, administered with either placebo or naloxone, a drug used to treat opiate overdose. A second goal is to determine if there are sex differences in these two drug regimens. Drugs will be administered with single-use intranasal spray devices. All participants will receive two sprays (one spray per nostril). One of the two sprays will be nalbuphine (5 mg). The other spray will be naloxone in half the participants and placebo in the other half.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of temporomandibular muscle pain OR
* Clinical diagnosis of burning mouth syndrome
* Pain duration: at least 3 months
* Pain severity: 2 or greater on a 0 - 10 scale

Exclusion Criteria:

* No adverse reaction to study drugs
* Not currently using narcotic analgesic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Levine, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment details unavailable due to death of investigator
Pre-assignment Details: pre-assignment details unavailable due to death of investigator
Groups:
- BMS Nalbuphine + Naloxone: nalbuphine plus naloxone : Patient group: burning mouth syndrome. Nalbuphine 5 mg administered by nasal spray (one time only). Naloxone 0.4 mg administered by nasal spray (one time only).
- BMS Nalbuphine + Placebo: nalbuphine plus placebo : Patient group: Burning mouth syndrome. Nalbuphine 5 mg administered by nasal spray (one time only). Placebo (naloxone vehicle) administered by nasal spray (one time only).
- TMD Nalbuphine + Naloxone: nalbuphine plus naloxone : Patient group: temporomandibular disorders. Nalbuphine 5 mg administered by nasal spray (one time only). Naloxone 0.4 mg administered by nasal spray (one time only).
- TMD Nalbuphine + Placebo: nalbuphine plus placebo : Patient group: temporomandibular disorders. Nalbuphine 5 mg administered by nasal spray (one time only). Placebo (naloxone vehicle) administered by nasal spray (one time only).
Period: Overall Study
Arm/Group | BMS Nalbuphine + Naloxone | BMS Nalbuphine + Placebo | TMD Nalbuphine + Naloxone | TMD Nalbuphine + Placebo
Started | 8 | 5 | 18 | 15
Completed | 8 | 5 | 18 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Co-investigators have spent many hours with computer-support personnel trying to locate data on the deceased investigators' computer, but could find nothing other than the gender and treatment assignment for 46 enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS Nalbuphine + Naloxone | BMS Nalbuphine + Placebo | TMD Nalbuphine + Naloxone | TMD Nalbuphine + Placebo | Total
Number analyzed (Participants) | 8 | 5 | 18 | 15 | 46
Age, Customized [Number; unit: Participants]
  Unknown | 8 | 5 | 18 | 15 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 15 | 13 | 38
  Male | 3 | 0 | 3 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 18 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity as Measured on a Visual Analogue Scale (VAS) Ranging From Zero to 100.
Time Frame: 20 minute intervals for three hours.
Population: as for baseline characteristics
Arm/Group | BMS Nalbuphine + Naloxone | BMS Nalbuphine + Placebo | TMD Nalbuphine + Naloxone | TMD Nalbuphine + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Dr. Robert Gear led this study and maintained data on his computer. Co-investigators have spent many hours trying to locate data on the deceased investigators' computer, but could find nothing other than minimal results data that did not include Adverse Event (AE)or SAE data.
Arm/Group | BMS Nalbuphine + Naloxone | BMS Nalbuphine + Placebo | TMD Nalbuphine + Naloxone | TMD Nalbuphine + Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Dr. Robert Gear led this study and maintained data on his computer. Co-investigators have spent many hours trying to locate data on the deceased investigators' computer, but could find nothing other than the minimal results data entered here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes